CLINICAL TRIAL: NCT00682838
Title: Improving Obstructive Sleep Apnea Management Via Wireless Telemonitoring
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 07-163; 080139 (Other: UCSD IRB)
Record Dates: First submitted 2008-05-12; First posted 2008-05-22 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Sleep Apnea Syndromes
Keywords: Treatment compliance; Self-management; Telemedicine
MeSH Terms: conditions — Sleep Apnea Syndromes; Patient Compliance | interventions — Self-Management

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Self-Management (SM) (Experimental): Active Intervention - Self-management: Self-management Educational component focused on sleep apnea and CPAP from a self-management perspective
  Interventions: Behavioral: Self-management
- Telemonitored Care (TC) (Active Comparator): Active Comparator - Telemonitored care: Telemonitored care Consists of CPAP therapist actively monitoring care at a distance, and acting on that data per a set protocol
  Interventions: Behavioral: Telemonitored care
- SM + TC (Experimental): Self-management and Telemonitored care: Combination of both SM + TC intervention
  Interventions: Behavioral: Self-management; Behavioral: Telemonitored care
- Usual care (UC) (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Self-management — Self-management
  Arms: SM + TC; Self-Management (SM)
Behavioral: Telemonitored care — Telemonitored care
  Arms: SM + TC; Telemonitored Care (TC)

SUMMARY:
Obstructive sleep apnea (OSA) is a major chronic condition affecting the quality of life of up to one-fifth of all Veterans. Because of disappointingly low adherence to the gold-standard treatment (continuous positive airway pressure therapy - CPAP), the Institute of Medicine has stated that new adherence strategies are needed that improve the quality of care, reduce social and economic costs, and help OSA patients live happier, healthier, and more productive lives through improved clinical management. The combination of a self-management approach along with emerging wireless technologies has strong potential to increase treatment adherence and improve outcomes.

DETAILED DESCRIPTION:
The Sleep Apnea Self-Management Program (SASMP) was evaluated by conducting a randomized, controlled trial of the program compared to Usual Care in patients diagnosed with OSA and prescribed CPAP therapy. Participants randomized to the SASMP group attended 4 weekly educational sessions of approximately two hours each. A trained leader facilitated the program from a scripted manual. Key topics covered in this program included: (1) management of OSA symptoms, CPAP side effects, and weight loss; (2) maintaining social contacts and family relationships; and (3) dealing with symptoms of depression and worries about the future.

The primary aim of this study was to examine the effect of the SASMP, compared to Usual Care, on CPAP adherence. It is hypothesized that SASMP participants will have higher levels of CPAP adherence compared to those in the Usual Care group.

A second aim of the study was to examine the effect of the SASMP, compared to Usual Care, on proposed mediating variables derived from social cognitive theory (perceived self-efficacy, outcome expectations). It is hypothesized that SASMP participants would have higher levels of self-efficacy and outcome expectations compared to the Usual Care group.

And the third aim of the study was to measure the short- and long-term effects of the SASMP, compared to Usual Care, on health outcomes (e.g., OSA symptoms and OSA-specific HRQOL). It is hypothesized that improvements in OSA symptoms and OSA-specific HRQOL will be seen both initially and as maintained 6 months and 1 year after the start of the SASMP.

ELIGIBILITY:
Inclusion criteria were:

1. Diagnosis of OSA
2. Prescription for CPAP treatment by a sleep physician
3. Being CPAP naïve (ie, no previous use of CPAP).

Exclusion criteria were:

1. Residence in a geographical area outside of San Diego County
2. Fatal comorbidity (life expectancy less than 6 months as indicated by treating physician)
3. Significant documented substance/chemical abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Management (SM): Active Intervention
  Self-management: Self-management Educational component focused on sleep apnea and CPAP from a self-management perspective
- Telemonitored Care (TC): Active Comparator
  Telemonitored care: Telemonitored care Consists of CPAP therapist actively monitoring care at a distance, and acting on that data per a set protocol
- SM + TC: 1+2
  Self-management: Self-management
  Telemonitored care: Telemonitored care
  Combination of both SM + TC intervention
- Usual Care: Usual care- control group
Period: Overall Study
Arm/Group | Self-Management (SM) | Telemonitored Care (TC) | SM + TC | Usual Care
Started | 65 | 67 | 75 | 73
Completed | 65 | 67 | 75 | 73
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The target population for this study is all Veterans with OSA. It was expected that most participants would be middle-aged and older men and women, from a variety of ethnic backgrounds and with a full range of medical co-morbidities.
Groups:
- Self-management: Active Intervention
  Self-management: Self-management
- Telemonitored Care: Active Comparator
  Telemonitored care: Telemonitored care
- SM+TC: 1+2
  Self-management: Self-management
  Telemonitored care: Telemonitored care
- Total: Total of all reporting groups
Arm/Group | Self-management | Telemonitored Care | SM+TC | Usual Care | Total
Number analyzed (Participants) | 65 | 67 | 75 | 73 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 57 | 66 | 62 | 241
  >=65 years | 9 | 10 | 9 | 11 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 3 | 9
  Male | 62 | 65 | 74 | 70 | 271
Region of Enrollment [Number; unit: participants]
  United States | 65 | 67 | 75 | 73 | 280

OUTCOME MEASURES:

1. Primary Outcome: Nightly CPAP Adherence
Description: Nightly CPAP adherence hours per night measured over the three-months period
Time Frame: 3 mos
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Self-management | Telemonitored Care | SM+TC | Usual Care
Number analyzed (Participants) | 65 | 67 | 75 | 73
hours per night | 3.7 (1.8) | 3.7 (2.3) | 3.7 (2.2) | 3.2 (2.3)
Statistical Analysis 1: Comparison: Self-management vs Telemonitored Care vs SM+TC vs Usual Care; Test type: Superiority or Other; p = 0.50, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Usual Care: Control Group
Arm/Group | Self-management | Telemonitored Care | SM+TC | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 0/75 | 0/73
Other Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 0/75 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes